CLINICAL TRIAL: NCT03794219
Title: Is Kinesio Taping Effective to the Radial Nerve in Patients With Lateral Epicondylitis? A Randomized-single Blind Study.
Brief Title: Is Kinesio Taping Effective to the Radial Nerve in Patients With Lateral Epicondylitis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Basak Mansiz-Kaplan, Principal Investigator of Department of Physical Medicine and Rehabilitation, Ankara Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E10654
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Athletic Tape; Naproxen

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio tape plus NSAID (Experimental): Kinesio tape is applied 3 times a week for 2 weeks with a total of 6 sessions in addition to 750 mg/day oral naproxen.
  Interventions: Other: Kinesio Tape; Drug: oral naproxen
- NSAID (Active Comparator): 750 mg/day oral naproxen is administered for 10 days.
  Interventions: Drug: oral naproxen

INTERVENTIONS:
Other: Kinesio Tape — To all patients,750 mg/day oral naproxen is administered for 10 days. Additionally, in intervention group kinesio tape is applied 3 times a week for 2 weeks with a total of 6 sessions.
  Arms: Kinesio tape plus NSAID
Drug: oral naproxen — 750 mg/day oral naproxen is administered for 10 days.

SUMMARY:
Lateral epicondylitis (LE) is the most frequent painful musculoskeletal condition, which is characterized by a pain in the lateral epicondyle of the humerus and the common extensor tendon. The incidence of LE is approximately one to three percent of general population. LE is mostly the result of the overuse and repetitive movements of wrists and hands because of occupational or recreational activities. Diagnosis depends on clinical symptoms, history and physical examination including manual provocation tests. Magnetic resonance imaging, ultrasound (US), x-ray and electrophysiological assessment may be used in patient who do not response to conservative treatments. It is known that the radial nerve cross sectional-areas (CSAs) are increased in cases of refractory LE, although nerve conduction studies are normal. There is insufficient evidence to prove the superiority of any of conservative treatments to the others in patients with LE. The literature indicates that Kinesio taping decreases pain intensity, recovers grip strength, and improves functional status in patients with LE. The investigators design a randomized, single-blind, controlled trail to evaluate the effects of Kinesio taping both clinical and using ultrasonography.

DETAILED DESCRIPTION:
After obtaining written informed consent, patients of clinically diagnosed with LE are randomized into intervention and control group. To all patients, activity modification is suggested and 750 mg/day oral naproxen is administered for 10 days. Additionally, in intervention group, kinesio tape was applied 3 times a week for 2 weeks with a total of 6 sessions. The primary outcome is visual analog scale (VAS) and secondary outcomes include the Patient-Rated Forearm Evaluation Questionnare (PRTEQ), CET thickness and radial nerve CSAs. The evaluation was performed pretreatment as well as on the 2nd week, and 6th week after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* the presence of pain in the lateral elbow region at least for three months
* tenderness around the lateral humeral epicondyle following at least one of these provocation tests: resisted wrist extension, resisted middle finger extension or passive stretch of wrist extensors.

Exclusion Criteria:

* bilateral LE
* presence of trigger point in the extensor muscles of the forearm
* history of proximal upper extremity or neck symptoms
* cervical pathology
* central or peripheral neurologic disease
* nerve entrapment syndromes
* surgical treatments for LE
* presence of condition that may prevent the patient using NSAIDs (i.e. gastrointestinal disorders, using anticoagulant)
* trauma history of upper extremity
* previous steroid injection around the lateral epicondyle
* physical therapy targeted for LE in the past 6 months
* presence of structures like fibrous bands, arc or recurrent radial artery around the radial nerve that may cause the entrapment of nerve
* pregnancy and having any systemic disease that may cause swelling at nerves such as diabetes mellitus, renal insufficiency, thyroid disease or rheumatic disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-07-07 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pain on 2nd and 6th weeks | Pre-treatment, 2nd and 6th weeks after treatment
  Using the Visual analog scale (VAS) to measure the pain scale before treatment and multiple time frame after treatment. The VAS is a straight horizontal line of fixed length, 10cm. The ends are defined as the extreme limits of the parameter to be measured orientated from the left (worst, 0) to the right (best, 10).

SECONDARY OUTCOMES:
Change from baseline of functional status on 2nd and 6th weeks | Pre-treatment, 2nd and 6th weeks after treatment
  Using Patient-Rated Forearm Evaluation Questionnare (PRTEQ) to evaluate functional status. The PRTEQ is a 15-item questionnaire which has two subscale: pain subscale and function subscale.. It is shown to be a reliable and valid tool for measuring pain and function in patients with LE. Pain subscale is comprised of 5 questions, and function subscale is comprised of 10 questions. The total score is calculated by the sum of these two subscales.
Change from baseline of common extensor tendon (CET) thickness on 2nd and 6th weeks | Pre-treatment, 2nd and 6th weeks after treatment.
  Using the musculoskeletal ultrasonography to measure CET thickness.
Change from baseline of radial nerve cross-sectional area (CSA) on 2nd and 6th weeks | Pre-treatment, 2nd and 6th weeks after treatment.
  Using the musculoskeletal ultrasonography to measure radial nerve cross-sectional area. Measurements of radial nerve CSA is taken from three different levels: spiral grove, just before bifurcation and between the two heads of supinator muscle (CSA)

CONTACTS AND LOCATIONS:
Locations (1):
- Basak Mansiz-Kaplan, Ankara, Turkey (Türkiye)